CLINICAL TRIAL: NCT04127396
Title: Exploring Lenvatinib Plus TACE Versus Sorafenib Plus TACE for Hepatocellular Carcinoma Patients With Portal Vein Tumor Thrombus: Efficacy, Safety and Outcome Analysis
Brief Title: Lenvatinib Plus TACE Versus Sorafenib Plus TACE for HCC With PVTT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Jinglong Chen, Chief of Oncology, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingDH 001
Record Dates: First submitted 2019-10-08; First posted 2019-10-15 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Carcinoma, Hepatocellular; Portal Vein Tumor Thrombus
Keywords: Transarterial chemoembolization; hepatocellular carcinoma; portal vein tumor thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lenvatinib and TACE (Experimental): Patients in Lenvatinib + TACE group will take oral lenvatinib within one day of randomization and receive TACE 1 day after oral administration of lenvatinib.
  Interventions: Drug: Lenvatinib Pill; Procedure: Transarterial chemoembolization(TACE)
- Sorafenib and TACE (Active Comparator): Patients in Sorafenib + TACE group will take oral sorafenib within one day of randomization and receive TACE 1 day after oral administration of lenvatinib.
  Interventions: Drug: Sorafenib; Procedure: Transarterial chemoembolization(TACE)

INTERVENTIONS:
Drug: Lenvatinib Pill — Lenvatinib capsules will be administered orally, once daily in continuous 28-day cycles. Body weight (BW)>60 kilograms(kg)-Lenvatinib 12 mg (taken as three 4-mg capsules); BW<60kg-Lenvatinib 8 mg (taken as two 4-mg capsules)
  Other Names: E7080
  Arms: lenvatinib and TACE
Procedure: Transarterial chemoembolization(TACE) — TACE will be performed one day after oral administration of lenvatinib . TACE with either cTACE or DEB-TACE can be used, depending on the condition of center.
  Arms: lenvatinib and TACE
Drug: Sorafenib — Sorafenib capsules will be administered orally, 400 mg twice daily (BID) oral dosing.
  Arms: Sorafenib and TACE
Procedure: Transarterial chemoembolization(TACE) — TACE will be performed one day after oral administration of Sorafenib. TACE with either cTACE or DEB-TACE can be used, depending on the condition of center.
  Arms: Sorafenib and TACE

SUMMARY:
Hepatocellular carcinoma (HCC) is the fourth most common cancer in China, with a crude incidence rate of 26.67 per 100,000 population. Moreover, 357,800 new liver cancer cases are predicted to be diagnosed in China in 2020. HCC represents approximately 90% of all cases of primary liver cancer. HCC has a high predilection for portal vein invasion, which occurs in 44-62% of living patients with HCC. Patients with PVTT usually have an aggressive disease course, decreased liver function reserve, limited treatment options, thus worse overall survival. Among untreated HCC patients with PVTT, the median overall survival has been reported as low as 2 to 4 months with supportive care. Sorafenib is the first-line treatment for HCC patients with PVTT, however, it has shown unsatisfactory benefit. Notably, sorafenib combined with TACE significantly improved the TTP over sorafenib alone, albeit for no more than 1 month in the median TTP, and the median OS was not significantly prolonged. A promising drug-lenvatinib was approved in China on September 2018, in the China patients subgroup analysis showed an encouraging results. Lenvatinib group had showed a significant benefit in TTP, PFS and ORR. Also median overall survival time was significantly improved in China subgroup (Lenvatinib group: 15 months VS Sorafenib group: 10.2 months). However, REFLECT didn't enrolled patients who had tumors invading the maint portal vein. The mechanisms of lenvatinib or sorafenib combined with TACE were still unknown, and clinical data were limited.

This study was to explore lenvatinib plus TACE versus sorafenib plus TACE for HCC with PVTT: efficacy and safety. Biomarkers expression of VEGFR, FGFR, FDGF-α, IL-2,etc would be detected to find the difference between the two groups, finally to analyze the relationship between clinical outcomes and biomarkers' expression. A better treatment modality to HCC with PVTT patients would be expected and promoted.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fourth most common cancer in China, with a crude incidence rate of 26.67 per 100,000 population. Moreover, 357,800 new liver cancer cases are predicted to be diagnosed in China in 2020, and HCC is by far the most common subtype of primary liver cancer and is the second most frequent cause of cancer-related death in the country. Approximately 80% of liver cancers are attributed to chronic infection with hepatitis B virus (HBV) and hepatitis C virus; other factors, including diabetes mellitus, non-alcoholic fatty liver disease, alcohol consumption, and tobacco use, have also been found to be potential risk factors for liver cancer HCC has a high predilection for portal vein invasion, which occurs in 44-62% of living patients with HCC. Portal vein tumour thrombosis (PVTT) usually portends a worse prognosis, with a median survival time of only 2.7-4.0 months in untreated patients. Despite advancements in understanding the molecular aetiology of HCC, the outcomes for patients with this disease who develop PVTT remain unsatisfactory.

Several treatment strategies for patients with inoperable HCC who developed PVTT have been attempted, including first-line targeted therapy with sorafenib, transarterial chemoembolisation (TACE), TACE plus sorafenib, percutaneous radiofrequency ablation (RFA), and radiotherapy. However, the prognosis of patients with HCC who are complicated by PVTT remains poor, and the optimal treatment modality for such patients has not been established to date.

Notably, sorafenib combined with TACE significantly improved the TTP over sorafenib alone, albeit for no more than 1 month; the median TTP was less than 3 months, and the median OS was not significantly prolonged.

In the recent phase III global multicentre REFLECT study, lenvatinib, the only other available first-line anti-angiogenic drug, did not improve overall survival (OS). However, lenvatinib as an oral multikinase inhibitor that targets VEGF receptors 1-3, FGF receptors 1-4, PDGF receptor α, RET and KIT, median time of PFS was 8.9 months (95% CI 7.4-9.2) for patients in the lenvatinib group compared to 3.7 months (95% CI 3.6-5.4) for patients in the sorafenib group. Lenvatinib also showed a greater objective response rate (ORR) than did sorafenib group. ORR was 40.6% (95% CI 36.2-45.0) for patients in the lenvatinib group compared to 12.4% (95% CI 9.4-15.4) for patients in the sorafenib group, and TTP was 7.4 (95% CI 7.2-9.1) VS 3.7 (95% CI 3.6-3.9). What's more, in the Chinese patients subgroup analysis showed an encouraging results, lenvatinib group not only showed significant improvement in PFS, TTP, ORR, but also in median OS time ( Lenvatinib group: 15 months VS sorafenib group 10.2 months). However, REFLECT didn't enrolled patients who had tumors invading the maint portal vein.

However, the mechanism of sorafenib combined with TACE was unknown, and clinical data of TACE plus lenvatinib for HCC had not been reported until now. As our preliminary experimental results showed that lenvatinib combined with TACE show a 91.7% clinical benefit in 11 cases HCC with PVTT (7 PR cases, 4 SD cases) , the median TTP was 6.5 months, during the preliminary experimental trail hadn't observed any fatal adverse event occurred.

In addition to these supporting data, lenvatinib plus TACE showed a potential benefit to HCC with PVTT patients. This study was to explore lenvatinib plus TACE versus sorafenib plus TACE for HCC with PVTT: efficacy and safety. Biomarkers expression of VEGFR, FGFR, PDGF-α, IL-2,etc would be detected to find the difference between the two groups, finally to analyze the relationship between clinical outcomes and biomarkers' expression.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically proven HCC.
2. HCC complicated by PVTT.
3. Patient had not received previous systemic therapy.
4. At least one measurable tumor along a single dimension according to the modified Response Evaluation Criteria in Solid Tumors (mRECIST).
5. WBC ≥ 3.0*109/L，PLT≥70*109/L，Hgb≥80*109/L；ALT≤2.5ULN，AST≤2.5ULN，TBIL≤3ULN，ALB≥28g/L；CCr ≥80ml/min.
6. Patients had not history of previous local therapy such as radiotherapy, hepatic arterial embolisation, chemoembolisation, RFA, percutaneous injection, or cryoablation.
7. Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 or 1;
8. Child-Pugh class A or Child-Pugh class B (score 7).
9. All patients were voluntary, and signed informed agreement.

Exclusion criteria

1. Previous or concomitant systemic therapy (including molecularly targeted therapies).
2. Known history of HIV infection.
3. Clinically serious infections.
4. Administered warfarin as an anticoagulant.
5. History of organ allograft.
6. History of cardiac disease.
7. Known central nervous system tumour.
8. Known gastrointestinal bleeding up to 30 days before study enrolment,
9. Pregnancy or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to progression | up to 18 months
  The primary endpoint was TTP (defined as the date of randomization until progression).
  Treatment response was evaluated according to mRECIST combined with contrast-enhanced dynamic CT or magnetic resonance imaging.

SECONDARY OUTCOMES:
Objective response rate(ORR) | up to 18 months
  ORR defined as the rate of patients with complete response or partial response according to mRECIST.
overall survival(OS) | up to 18 months
  OS defined as the date of randomization to death from any cause.
adverse events(AEs) | up to 18 months
  AEs(adverse events) evaluated by the CTC-AE 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding X, Sun W, Li W, Shen Y, Guo X, Teng Y, Liu X, Zheng L, Li W, Chen J. Transarterial chemoembolization plus lenvatinib versus transarterial chemoembolization plus sorafenib as first-line treatment for hepatocellular carcinoma with portal vein tumor thrombus: A prospective randomized study. Cancer. 2021 Oct 15;127(20):3782-3793. doi: 10.1002/cncr.33677. Epub 2021 Jul 8. PMID 34237154